CLINICAL TRIAL: NCT06574594
Title: Effect of Methotrexate Discontinuation on Immunogenicity of Shingrix in Patients With Rheumatoid Arthritis
Brief Title: Effect of MTX Discontinuation on Shingrix Response in RA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Hong Ki Min, Assistant Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-02-038
Record Dates: First submitted 2024-08-21; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis
Keywords: herpes zoster; Shingrix; methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid; Herpes Zoster | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTX discontinuation (Experimental): methotrexate stop for 2 weeks after each shingrix vaccination
  Interventions: Drug: Methotrexate
- MTX continuation (Active Comparator)
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — methotrexate discontinuation group : stop MTX for 2 weeks after each shingrix vaccination
  Arms: MTX discontinuation
Drug: Methotrexate — methotrexate continuation group : keep methotrexate
  Arms: MTX continuation

SUMMARY:
The goal of this clinical trial is to learn if methotrexate discontinuation affect on immunogeneity of shingrix in RA patients. The main questions it aims to answer are:

Discontinuation of methotrexate after shingrix immunization increase efficacy of the vaccine in patients with RA ?

Researchers will compare humoral and cell-mediated immunity against herpes zoster in RA patients who are vaccinated by shingrix, and compare these immunity between RA patients with MTX discontinuation and MTX continuation groups.

Participants will:

Vaccinated with shingrix twice. MTX continuation group will keep taking MTX after shingrix vaccination, whereas MTX discontinuation group will stop MTX for 2 weeks after shingrix vaccination.

Visit the clinic at baseline (first shingrix vaccination), 2 months later for 2nd shingrix vaccination, then 3 & 6 months later from baseline to achieve blood sample.

ELIGIBILITY:
Inclusion Criteria:

* fulfill 2010 ACR/EULAR classification criteria for rheumatoid arthritis
* age over 19 years
* methotrexate user
* agree for vaccination with shingrix

Exclusion Criteria:

* have other form of inflammatory arthritis or autoimmune-mediated disease
* malignancy, current infection, pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-08-22 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cell-mediated immunity (CD4+ and CD8+ T cell against herpes zoster) | baseline (before 1st vaccination), 1 months later from 2nd vaccination, 3 months later from 2nd vaccination

SECONDARY OUTCOMES:
, Humoral immunity (anti-VZV antibody, anti-gE antibody) | baseline (before 1st vaccination), 1 months later from 2nd vaccination, 3 months later from 2nd vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ki Min, MD, PhD, Study Chair — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD can be shared with reasonable request.